CLINICAL TRIAL: NCT05200871
Title: Humanistic Burden of Rare Kidney Diseases: Understanding the Impact of FSGS and IgAN on Patients and Caregivers Study (HONUS) - A Multi-National, Cross-Sectional Survey Study
Brief Title: Humanistic Burden of (FSGS) Focal Segmental Glomerulosclerosis and IgAN (Immunoglobulin A Nephropathy)
Acronym: HONUS
Status: Completed | Type: Observational
Sponsor: Travere Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: TVTX-RE021-402
Record Dates: First submitted 2021-11-22; First posted 2022-01-21 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Focal Segmental Glomerulosclerosis; Immunoglobulin A Nephropathy
Keywords: Observational; Cross-Sectional; Survey; Health-related quality of life (HRQoL); Patients; Care-Partners; Humanistic; Burden
MeSH Terms: conditions — Glomerulosclerosis, Focal Segmental; Glomerulonephritis, IGA

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Adult patients: Adult patients (at least 18 years old) with FSGS or IgAN located in each of the six countries
- Adult patient care-partners of adult patients: Adult care-partners (paired with adult patients) (at least 18 years old) of adult patients with FSGS or IgAN located in each of the six countries
- Adult patient care-partners of pediatric/adolescent patients: Adult parents/care-partners (paired with adult patients) (at least 18 years old) of pediatric/ adolescent patients with FSGS or IgAN located in each of the six countries

SUMMARY:
The aim of this observational study is to assess humanistic burden among adults and children/adolescents with FSGS and IgAN as well as the burden and impact for patient care-partners in six countries (United States [US], United Kingdom [UK], France, Germany, Italy and Spain).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients and their adult care-partners: At least 18 years old; Either have a physician-provided diagnosis of FSGS or IgAN (with renal biopsy confirmation of the diagnosis) or being a care-partner for someone with a physician-provided diagnosis of FSGS or IgAN (with renal biopsy confirmation of the diagnosis);
* Able to provide informed consent;
* Located in the United States (US), United Kingdom (UK), Germany, France, Spain or Italy.

  *Care-partners (paired with adult patients) (defined as the individual [e.g., spouse, parent, sibling, relative, or friend] providing direct disease-related support to the adult patient.

  **All patient groups including chronic kidney disease (CKD) stage 1-5, with or without dialysis, and with or without kidney transplant will be included.
* Care-partners/parents of children/adolescents: At least 18 years old;
* Being a care-partner of children/adolescents with physician-provided diagnosis of FSGS or IgAN (with renal biopsy or genetic confirmation of the diagnosis);
* Able to provide informed consent; Located in the US, UK, Germany, France, Spain or Italy.

  * Care-partners will be defined as family members who provide disease-related support and unpaid care to child/adolescent patients

Exclusion Criteria:

* Patient has FSGS or IgAN secondary to another condition;
* Patient has a history of malignancy other than adequately treated basal cell or squamous cell skin cancer;
* Patient has a co-existing glomerular disease (e.g., membranous nephropathy, lupus nephritis);
* Patient is currently participating in a kidney disease clinical trial, and potentially receiving active treatment as part of the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include adult patients with FSGS or IgAN and their adult care-partners, as well as parents/care-partners of children/adolescents with FSGS or IgAN, who meet specified inclusion/exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 487 (Actual)
Dates: Start 2022-02-05 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Demographics | Day 1, day of enrollment
  Adult patients (self-reported) - age, sex, education level, household income, marital status, current work status, race/ethnicity (for patients in the US and in the UK), health insurance (for patients in the US), approximate travel time to receive FSGS/IgAN medical care.
  Child/adolescent patients (reported by parent/care-partner) - age, sex, current school status, race/ethnicity (for patients in the US and in the UK), approximate travel time to receive FSGS/IgAN medical care.
  Care-partners of adult patients and parents/care-partners of child/adolescent patients - age, sex, education level, household income, marital status, relationship to person with FSGS/IgAN, current work status, race/ethnicity (for patients in the US and UK).
Disease history. | Day 1, day of enrollment
  Adult patients (self-reported) - length of time from onset of symptoms to diagnosis, time since diagnosis, renal biopsy status, comorbidities, CKD (Chronic kidney disease) stage at diagnosis, current CKD stage (including dialysis status), transplant status (including type of transplant and occurrence of rejection or recurrence of disease), current level of proteinuria.
  Pediatric/adolescent patients (reported by parent/care-partner) - length of time from onset of symptoms to diagnosis, time since diagnosis, renal biopsy status, comorbidities, CKD stage at diagnosis, current CKD stage (including dialysis status), transplant status (including type of transplant and occurrence of rejection or recurrence of disease), current level of proteinuria.
Adult patient health-related quality of life. | Day 1, day of enrollment
  Measured by Kidney Disease Quality of Life 36-item Short Form Survey (KDQOL-36).
Pediatric patient health-related quality of life (reported by parent/care-partner). | Day 1, day of enrollment
  Measured by Pediatric Quality of Life Inventory (PedsQL) Parent report for teens (ages 13-18) or Parent report for children (ages 8-12).
Adult patient care-partner and pediatric patient parent/care-partner health-related quality of life. | Day 1, day of enrollment
  Measured by 12-Item Short Form Health Survey (SF-12).
Adult patient, adult patient care-partner and pediatric patient parent/care-partner anxiety. | Day 1, day of enrollment
  Measured by General Anxiety Disorder 7 (GAD-7) questionnaire.
Adult patient, adult patient care-partner and pediatric patient parent/care-partner depression. | Day 1, day of enrollment
  Measured by Patient Health Questionnaire 9 (PHQ-9) module.
Adult patient cognition. | Day 1, day of enrollment
  Measured by cognition items of the Massachusetts General Hospital (MGH) Cognitive and Physical Functioning Questionnaire (CPFQ).
Adult patient symptoms. | Day 1, day of enrollment
  Measured by 5-point Likert scale ranking of most burdensome symptoms.
Pediatric patient symptoms (reported by parent/care-partner). | Day 1, day of enrollment
  Measured by 5-point Likert scale ranking of most burdensome symptoms.
Adult patient, pediatric patient (reported by parent/care-partner), adult patient care-partner and pediatric patient parent/care-partner fear and anxiety for the future. | Day 1, day of enrollment
  Measured by 5-point Likert scale fear and anxiety for the future.
Adult patient productivity impairment. | Day 1, day of enrollment
  Measured by Work Productivity and Activity Impairment Questionnaire: Specific Health Problem (WPAI:SHP).
Adult patient care-partner and pediatric patient parent/care-partner productivity impairment. | Day 1, day of enrollment
  Measured by Work Productivity and Activity Impairment Questionnaire (WPAI) caregiver version.
Adult patient, adult patient care-partner and pediatric patient parent/care-partner impact of disease. | Day 1, day of enrollment
  Measured by and 5-point Likert scale impact on education, career, employment, relationships, personal finances and lifestyle.
Pediatric/adolescent patient impact of disease (reported by parent/care-partner). | Day 1, day of enrollment
  Measured by 5-point Likert scale impact on patient education, career (adolescents), employment (adolescents), relationships and lifestyle.

CONTACTS AND LOCATIONS:
Overall Officials: Leah Conley, MBA, Study Director — Travere Therapeutics
Locations (6):
- United States (4):
  - Travere Investigational Site, San Francisco, California
  - Travere Investigational Site, Belmar, New Jersey
  - Travere Investigational Site, Chapel Hill, North Carolina
  - Travere Investigational Site, King of Prussia, Pennsylvania
- Travere Investigational Site, Villingen-Schwenningen, Germany
- Travere Investigational Site, Madrid, Spain